CLINICAL TRIAL: NCT04924998
Title: Clinical Study Protocol for the Treatment of Immunoglobulin Light Chain Amyloidosis Cardiomyopathy
Brief Title: Clinical Study for AL-CM
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0133
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Immunoglobulin Light Amyloidosis Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AL-CM
  Interventions: Drug: current treatment of AL-CM

INTERVENTIONS:
Drug: current treatment of AL-CM — current treatment of AL-CM

SUMMARY:
In this study, patients diagnosed with Al-CM were selected to observe the effect of treatment and conduct long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 years, regardless of gender, diagnosed with Al-CM at the Second Affiliated Hospital of Zhejiang University School of Medicine;
* Patients have the ability to understand the test, can cooperate with investigators.

Exclusion Criteria:

* Unable to understand or unwilling to fill in informed consent forms or follow visitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AL-CM
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 10 year
  incidences of MACE-4(cardiovascular death, myocardial infarction, stroke and hospitalized unstable angina)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China